CLINICAL TRIAL: NCT02591251
Title: A Comparison Between Povidone-iodine and Normal Saline Solution in Preoperative Vaginal Cleansing in Laparoscopic Surgery: a Randomized Clinical Study
Brief Title: Povidone-iodine Versus Normal Saline Solution in Vaginal Cleansing in Laparoscopy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: VCL
Record Dates: First submitted 2015-10-28; First posted 2015-10-29 (Estimated); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Postoperative Infection
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- The povidone-iodine group (Active Comparator): The patients will be subjected to povidone-iodine (Betadine7.5%, Phama Care) for vaginal cleaning before the laparoscopic surgery
  Interventions: Drug: Povidone-iodine solution
- Normal saline group (Active Comparator): The patients will be subjected to normal saline solution (Sod. Chloride 0.9%, Nile) for vaginal cleaning before the laparoscopic surgery.
  Interventions: Drug: Normal saline solution

INTERVENTIONS:
Drug: Povidone-iodine solution
  Arms: The povidone-iodine group
Drug: Normal saline solution
  Arms: Normal saline group

SUMMARY:
Laparoscopy is a minimally invasive method used for diagnostic and therapeutic purposes. It allows surgeons to take a look on the abdominal and pelvic organs. Diagnostic laparoscopy is usually done in an operating room under general anesthesia. The procedure takes about 25 minutes and the patients usually discharged in the same day. The laparoscopy can diagnose pelvic pathological conditions in approximately 50% of the cases. However, the laparoscopy has some complications, such as infections, hemorrhage and injuries of visceral organs.

A preoperative vaginal preparation is important to prevent the bacteria colonization in a trial to avoid postoperative infection after laparoscopic surgery. The povidone-iodine (PI) is normally used as a skin and vaginal disinfectant to prevent postoperative infections, however; it can be the cause of significant postoperative irritation.

There are many reports in the literature proved that the mechanical cleansing of the vagina, not the use of an antiseptic solution, is responsible for the efficacy of vaginal preparations. In the field of assisted reproductive technology; A study in 1992 concluded that the infection rates with normal saline solution are comparable to PI.

Another proved that, a normal saline solution can be effective in prevention of preventing postoperative infections after vaginal surgery.

The most recent study by Lewis et al has been shown that the Baby shampoo is preferable than PI in vaginal cleansing before gynecologic procedures because it has minimal vaginal irritation and cheaper than PI.

So the optimal vaginal antiseptic solution is unknown, the investigators want to conduct a randomized trial comparing 2 commonly used vaginal antiseptic solutions: PI and the saline solution before the laparoscopic surgery.

The normal saline is used in medicine as an intravenous isotonic infusion and for cleaning wounds. It is a mild but effective cleaning agent and will not harm normal tissue, unlike many stronger antiseptics. It is available and inexpensive in comparison to povidone iodine.

ELIGIBILITY:
Inclusion Criteria:

1 - All women who will subject to laparoscopy (diagnostic or operative) for gynecological problems

Exclusion Criteria:

1 - All women who will subjected to operative laparoscopy for myomectomy or hysterectomy.

2- All patients have current vaginitis or urinary tract infection before the laparoscopy.

3- Diabetic women. 4- Women with BMI > 25 kg/m2.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2015-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Degree of fever postoperative (c) | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No